CLINICAL TRIAL: NCT03602664
Title: Postoperative Recovery and Longterm Outcome After Thoracic Surgery
Brief Title: Postoperative Recovery After Thoracic Surgery
Acronym: POLO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Stefan Lundin, Adj Professor, Sahlgrenska University Hospital
Other Study IDs: LUA-74206
Record Dates: First submitted 2018-06-05; First posted 2018-07-27 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Postoperative Pain; Postoperative Complications
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Thoracic surgery: Patients undergoing thoracic surgery

SUMMARY:
A questionaire specifically developed using in depth interviews with patients that has undergone surgery has been developed. This questionaire will be used for longterm follow in patients undergoing thoracic surgery. 200 patients will be asked to fill in this questionaire preoperatively as well as 3 and 12 months after surgery to assess symptomburden after surgery with specific aim to study postoperative pain as well as other physical, mental and cognitive problems that may affect the patient and their daily activities, health, return to work, family life and economy.

DETAILED DESCRIPTION:
In Sweden around 400 000 patients under go surgical operations in hospitals. A large proportion, around 20%, develop persistent postoperative pain which affects their quality of life and their recovery towards a normal life.

A questionaire specifically developed using in depth interviews with patients that has undergone surgery has been developed. This questionaire will be used for longterm follow in patients undergoing thoracic surgery. 200 patients will be asked to fill in this questionaire preoperatively as well as 3 and 12 months after surgery to assess symptomburden after surgery with specific aim to study postoperative pain as well as other physical, mental and cognitive problems that may affect the patient and their daily activities, health, return to work, family life and economy.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing thoracic surgery (thoracotomy or thoracoscopy) who accept to participate in the study

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients planned to undergo thoracotomy or thoracoscopy at Sahgrenska University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-06-05 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain 3 months after surgery as compared to preoperatively assessed with a studyspecific questionnaire | Pain at 3 months after surgery as compared to preoperatively
  Pain at 3 months after surgery as compared to prior to surgery

SECONDARY OUTCOMES:
Postoperative functional impairment after surgery assessed with a studyspecific questionnaire | Status at 3 months after surgery as compared to before the operation
  Physical, mental and cognitive problems were assessed with a studyspecific questionaire 3 months after surgery as compared to preoperatively
Postoperative functional impairment 12 months after surgery assessed with a studyspecific questionnaire 12 month after surgery | Status 12 months after surgery compared to before surgery
  Physical, mental and cognitive problems 12 months after surgery
Postoperative pain 12 months after surgery as compared to preoperatively assessed with a studyspecific questionnaire | Pain at 12 months after surgery as compared to preoperatively
  Pain at 12 months after surgery as compared to prior to surgery

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Lundin, MD PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No